CLINICAL TRIAL: NCT05579158
Title: Effects of Time-restricted Eating Supported by Mobile Technology in Patients With Non-alcoholic Fatty Liver Disease: Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University (Other)
Collaborators: National Institute of Health, Korea (Other Government)
Responsible Party: Principal Investigator, Dae Won Jun, Professor, Hanyang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HanyangU
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Time Restricted Feeding; Mobile Technology
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Intermittent Fasting | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mobile application-supported both calorie restriction and time-restricted eating (mCR/TRE) (Experimental): This arm receives wearable device and mobile application-supported nutritional counseling for four months. The nutritional counseling consists of both calorie restriction (500kcal below estimated energy requirement) and time-restricted eating (an 8-hour period (from 10 a.m. to 6 p.m.) each day).
  Interventions: Behavioral: Mobile application and wearable device; Behavioral: Time-restricted eating
- Mobile application-supported calorie restriction (mCR) (Active Comparator): This arm receives wearable device and mobile application-supported nutritional counseling for four months. The nutritional counseling consists of only calorie restriction (500kcal below estimated energy requirement).
  Interventions: Behavioral: Mobile application and wearable device
- Calorie restriction (CR) (No Intervention): Standard of care. This arm receives a brief counseling of calorie restriction.

INTERVENTIONS:
Behavioral: Mobile application and wearable device — Mobile application-supported nutritional counseling includes education, monitoring, interaction, and physical activity
  Arms: Mobile application-supported both calorie restriction and time-restricted eating (mCR/TRE); Mobile application-supported calorie restriction (mCR)
Behavioral: Time-restricted eating — Time-restricted eating (an 8-hour period (from 10 a.m. to 6 p.m.) each day)
  Arms: Mobile application-supported both calorie restriction and time-restricted eating (mCR/TRE)

SUMMARY:
In non-alcoholic fatty liver disease (NAFLD), it is established that calorie restriction is the most essential dietary modification. The time-restricted diet is successful lowering total calorie consumption and insulin resistance, and is anticipated to be beneficial for patients with NAFLD. Therefore, this study aims to conduct a prospective study to determine the effect of time-restricted diet via a mobile application on the amount of intrahepatic fat and 10-year cardiovascular disease risk in patients with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 19 years who are willing and able to complete all procedures
* Hepatic steatosis by imaging (ultrasound, computed tomography, magnetic resonance imaging, and controlled attenuation parameter (≥260 dB/m))

Exclusion Criteria:

* Body mass index (BMI) <23
* Other causes of chronic liver disease (HBV, HCV), autoimmune diseases or chronic cholestatic liver disease
* Medications which cause liver disease or secondary hepatic steatosis (Tamoxifen, systemic corticosteroids, methotrexate, tetracycline, estrogens, valproic acid, and statin (registration is possible if statin is delivered in a consistent dosage within 12 weeks)
* Significant alcohol intake (>210g/week for men, >140g/week for women)
* Severe medical comorbidities (ischemic heart disease, 3rd degree atrioventricular block, chronic obstructive pulmonary disease, severe hypertension (blood pressure > 200/120 mmHg)
* Psychiatric illnesses which limit ability to exercise safely
* Diagnosed with diabetes on medication or insulin
* Participation in a weight-loss program within 12 weeks
* MRI contraindications

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Change in hepatic steatosis (%) | 16 weeks
  Change in hepatic steatosis (%) on Magnetic Resonance Imaging (MRI) Proton Density Fat fraction (PDFF) of the Liver

SECONDARY OUTCOMES:
Change in 10-year atherosclerotic cardiovascular disease (ASCVD) risk | 16 weeks
  Evaluate the mean change in atherosclerotic cardiovascular disease (ASCVD) risk score (%) (high ASCVD risk score means high risk of ASCVD)
Change in liver fibrosis (kPa) by Magnetic Resonance Elastography (MRE) | 16 weeks
  Evaluate the mean change in liver fibrosis (kPa) on Magnetic Resonance Elastography (MRE) of the Liver
Change in body weight (kg) | 16 weeks
  Evaluate the mean change in body weight (kg)
Change in systolic blood pressure (mmHg) | 16 weeks
  Evaluate the mean change in systolic blood pressure (mmHg)
Change in low-density lipoprotein level (mg/dL) | 16 weeks
  Evaluate the mean change in low-density lipoprotein level (mg/dL)
Change in serum alanine aminotransferase level (IU/L) | 16 weeks
  Evaluate the mean change in serum alanine aminotransferase level (IU/L)
Change in hemoglobin A1c level (%) | 16 weeks
  Evaluate the mean change in hemoglobin A1c level (%)
Change in insulin sensitivity | 16 weeks
  Evaluate the mean change in homeostatic model assessment for insulin resistance (HOMA-IR)
Change in urine microalbumin (mcg/min) | 16 weeks
  Evaluate the mean change in urine microalbumin (mcg/min)
Change in body muscle mass (kg) | 16 weeks
  Evaluate the mean change in body muscle mass (kg) as measured by bioelectrical impedance analysis (InBody)
Change in liver fibrosis by liver stiffness (kPa) | 16 weeks
  Evaluate the mean change in liver fibrosis by liver stiffness (kPa) under FibroScan®
Change in liver steatosis by controlled attenuation parameter (dB/m) | 16 weeks
  Evaluate the mean change in liver steatosis by controlled attenuation parameter (dB/m) under FibroScan®
Change in body weight (kg) at 6 months after the intervention | 40 weeks
  Evaluate the mean change in body weight (kg) at 24 weeks after the end of 16-week intervention period
Change in body weight (kg) at 12 months after the intervention | 64 weeks
  Evaluate the mean change in body weight (kg) at 48 weeks after the end of 16-week intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Dae Won Jun, M.D., Ph.D., Study Chair — Hanyang University
Locations (1):
- Hanyang University Seoul Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oh JH, Yoon EL, Park H, Lee S, Jo AJ, Cho S, Kwon E, Nah EH, Lee JH, Park JH, Ahn SB, Jun DW. Efficacy and safety of time-restricted eating in metabolic dysfunction-associated steatotic liver disease. J Hepatol. 2025 Dec;83(6):1256-1265. doi: 10.1016/j.jhep.2025.06.005. Epub 2025 Jun 19. PMID 40543603